CLINICAL TRIAL: NCT02619461
Title: The Acute Effect of High Intensity Exercise on Appetite, Appetite-regulating Hormones, and Bio-markers of Inflammation and Stress in Lean and Obese Boys
Brief Title: The Acute Effect of Exercise on Appetite Appetite-regulating Hormones and Inflammation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Study Investigator, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HIT_Exercise_Appetite_001
Record Dates: First submitted 2015-05-27; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Exercise at 70%VO2max on a recumbent bicycle for 30 minutes.
  Interventions: Other: Exercise
- Control (No Intervention): Resting

INTERVENTIONS:
Other: Exercise — Exercise at 70%VO2max on a recumbent bicycle for 30 minutes to investigate the effects of exercise at high intensities on appetite and biomarkers of appetite and inflammation.
  Arms: Exercise

SUMMARY:
This study describes the effect of acute high intensity exercise at 70% VO2peak on inflammation, stress, appetite hormones and appetite in lean and obese children and adolescents.

DETAILED DESCRIPTION:
In summary, exercise does induce a variety of metabolic mechanisms on a central and peripheral level, related to appetite other than solely gut peptides. The literature points towards a rather loose coupling when it comes to high intensity exercise and the suppression of food intake, without a clear explanation of the cause of exercise induced anorexia. This study is aimed to investigate high-intensity exercise and its effects on appetite and satiety hormones, inflammation, stress and eating behaviors on appetite and food intake.

The objective of the current study is to investigate the factors contributing to exercise-induced anorexia in lean and obese children, and maximize its translation into post-exercise suppression of food intake and promotion of negative energy balance particularly in obese children. It is hypothesized that high-intensity exercise would promote a greater suppression of food intake through suppression of appetite ratings via physiological mechanisms depending on stress and inflammation rather than gut peptides.

ELIGIBILITY:
Inclusion Criteria:

* 11 normal weight and 11 obese boys will be recruited for the study. Lean and obese boys aged 10-18 years, born full-term and with a normal body weight at birth, will be included in the study

Exclusion Criteria:

* Dieters and individuals with lactose intolerance, allergies to milk and dairy products and gastrointestinal problems will be excluded from the study.

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Appetite as assessed via visual analog scales | Timeperiod of 2 hours during each study intervention.
  Appetite will be assessed via visual analog scales. Each item will be scored from 0-100; 0 not hungry; 100 very hungry
Biomarkers of appetite | 4 timpoints during 2 hours during each study intervention.
  Biomarkers of appetite will be assessed such as A. Ghrelin; GLP-1; PYY and Leptin
Biomarkers of Inflammation | 4 timpoints during 2 hours during each study intervention.
  Biomarkers of inflammation will be assessed such as IL-6; IL-1beta; TNF-alpha; CRP

SECONDARY OUTCOMES:
Biomarkers of Stress | 4 timpoints during 2 hours during each study intervention.
  Biomarkers of stress will be assessed such as Cortisol and Adrenalin

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hunschede S, El Khoury D, Antoine-Jonville S, Smith C, Thomas S, Anderson GH. Acute changes in substrate oxidation do not affect short-term food intake in healthy boys and men. Appl Physiol Nutr Metab. 2015 Feb;40(2):168-77. doi: 10.1139/apnm-2014-0188. Epub 2014 Oct 22. PMID 25603432
- [Background] Tamam S, Bellissimo N, Patel BP, Thomas SG, Anderson GH. Overweight and obese boys reduce food intake in response to a glucose drink but fail to increase intake in response to exercise of short duration. Appl Physiol Nutr Metab. 2012 Jun;37(3):520-9. doi: 10.1139/h2012-038. Epub 2012 Apr 25. PMID 22530879
- [Background] Bozinovski NC, Bellissimo N, Thomas SG, Pencharz PB, Goode RC, Anderson GH. The effect of duration of exercise at the ventilation threshold on subjective appetite and short-term food intake in 9 to 14 year old boys and girls. Int J Behav Nutr Phys Act. 2009 Oct 9;6:66. doi: 10.1186/1479-5868-6-66. PMID 19818131
- [Derived] Hunschede S, Kubant R, Akilen R, Thomas S, Anderson GH. Decreased Appetite after High-Intensity Exercise Correlates with Increased Plasma Interleukin-6 in Normal-Weight and Overweight/Obese Boys. Curr Dev Nutr. 2017 Feb 28;1(3):e000398. doi: 10.3945/cdn.116.000398. eCollection 2017 Mar. PMID 29955695